CLINICAL TRIAL: NCT06286683
Title: Impact of Early Out-of-bed Mobilization on Physiological Parameters of Patients Admitted to Intensive Care for Subarachnoid Hemorrhage
Brief Title: Impact of Early Mobilization on SAH Patients Physiological Parameters
Acronym: MOBALPAH
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231706
Record Dates: First submitted 2024-02-14; First posted 2024-02-29 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Early mobilization; Brain perfusion; Transcranial doppler; Near-infrared spectroscopy; Lung Ultrasound
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Ultrasonography, Doppler, Transcranial; Spectroscopy, Near-Infrared; Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to intensive care: Patients admitted to intensive care for aneurysmal subarachnoid hemorrhage (SAH) and eligible for their first out-of-bed mobilization
  Interventions: Device: lung ultrasound; Device: Transcranial Doppler; Device: near-infrared spectroscopy (NIRS); Device: clinical examination

INTERVENTIONS:
Device: lung ultrasound — Used to diagnose and monitor pulmonary aeration in the context of prolonged decubitus disorders (atelectasis) via the lung ultrasound score (LUS).
Device: Transcranial Doppler — Non-invasive, bedside method of measuring cerebral blood flow.
Device: near-infrared spectroscopy (NIRS) — Non-invasive, bedside method of cerebral oximetry that requires no advanced expertise.
Device: clinical examination — clinical examination

SUMMARY:
The aim of the study is to evaluate the physiological response to out-of-bed mobilization in patients admitted to the intensive care unit for subarachnoid hemorrhage. More specifically, the aim is to measure the impact on cerebral perfusion, lung aeration, cardiovascular and respiratory parameters.

DETAILED DESCRIPTION:
In patients with subarachnoid hemorrhage, the mobilization strategy has been little studied. Several studies have already evaluated the consequences of mobilization in bed. Because of the deleterious consequences of prolonged bed rest, and in line with recommendations, practices have evolved towards early out-of-bed mobilization, which has shown benefits. However, the physiological consequences of out-of-bed mobilization have not yet been assessed. The aim of this study is to measure the impact of early out-of-bed mobilization of patients admitted for SAH on neuro-cardio-pulmonary physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

* Aneurysmal SAH
* Severity score World Federation Neurological Surgeons I to IV
* Secured aneurysm
* Eligible for their first early mobilization

Exclusion Criteria:

* Sedated patient
* Disturbed alertness, coma
* Unsecured aneurysm
* Patients under legal protection (guardianship, curatorship, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to intensive care for aneurysmal subarachnoid hemorrhage (SAH) and eligible for their first outof-bed mobilization
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Impact on lung aeration | at T0 before initiation of out-of-bed mobilization, and 15 minutes after moving to the chair.
  Lung Ultrasound Score by lung ultrasound, Ranging from 0 (normal lungs) to 36 (worst case scenario).

SECONDARY OUTCOMES:
Impact on cerebral blood flow | At T0 before initiation of out-of-bed mobilization, immediately after moving to the edge the bed, immediately after moving to the chair.
  cerebral blood flow using average velocities on transcranial Doppler
Impact on cerebral tissue oxygenation | At T0 before initiation of out-of-bed mobilization, immediately after moving to the edge the bed, immediately after moving to the chair.
  cerebral tissue oxygenation via NIRS
Impact on heart rate | At T0 before initiation of out-of-bed mobilization, immediately after moving to the edge the bed, immediately after moving to the chair.
  Heart rate
Impact on arterial pressure | At T0 before initiation of out-of-bed mobilization, immediately after moving to the edge the bed, immediately after moving to the chair.
  Arterial pressure
Impact on Saturation | At T0 before initiation of out-of-bed mobilization, immediately after moving to the edge the bed, immediately after moving to the chair.
  Saturation
Impact on neurological examination | At T0 before initiation of out-of-bed mobilization, immediately after moving to the edge the bed, immediately after moving to the chair.
  Glasgow Coma Scale score (scored between 3 and 15, 3 being the worst and 15 the best)
Impact on patient comfort | At T0 before initiation of out-of-bed mobilization, immediately after moving to the edge the bed, immediately after moving to the chair.
  Numerical Pain Rating Scale (scored between 0 and 10, 0 being "no pain",10 "the worst pain imaginable")

CONTACTS AND LOCATIONS:
Locations (1):
- Adéla FOUDHAÏLI, Paris, France

IPD SHARING:
Plan to Share IPD: No